CLINICAL TRIAL: NCT01558154
Title: Comparison of Treatment Effect of Chinese Medicine and Western Medicine on Depression in China and America
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: California Pacific Medical Center Research Institute (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Xue Yan, Psychology Department, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2011DFA30960
Record Dates: First submitted 2012-03-02; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Depression
Keywords: depression; Chinese herb; acupuncture; Psychotherapy; Transcranial magnetic stimulation
MeSH Terms: conditions — Depression | interventions — Acupuncture Therapy; Psychotherapy; Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Chinese herb (Experimental): Chinese herbs special for depression
  Interventions: Drug: Chinese herbs
- acupuncture (Experimental)
  Interventions: Procedure: acupuncture
- Psychotherapy (Experimental)
  Interventions: Other: Psychotherapy
- physiotherapy (Experimental)
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Drug: Chinese herbs — Chinese herbs special for depression
  Arms: Chinese herb
Procedure: acupuncture — six acupuncture point including DU20, EX HN3, EX HN1, PC6,HT7,SP6,special for depression
  Arms: acupuncture
Other: Psychotherapy — Thought Imprint Psychotherapy under lower Resistance State
  Arms: Psychotherapy
Device: Transcranial magnetic stimulation — Give magnetic stimulation at head
  Arms: physiotherapy

SUMMARY:
Comparison of different assessment methods to evaluate the treatment efficacy of Chinese medicine on minor and mild depression.

DETAILED DESCRIPTION:
Significant differences show on the evaluation of treatment efficacy of Chinese medicine on depression in China and America. Choose minor and mild depression patients as trials. One hundred and sixty trials will be included and randomly divided into Chinese medicine group (n=40), acupuncture group (n=40), traditional Chinese medicine psychology group (n=40) and physical treatment group (n=40). Time points of assessment are before treatment, 1 week, 2 weeks, 4weeks, 6 weeks and 12 weeks post treatment.The assessment tools are series of psychological questionnaires. And study the mechanism of treatment efficacy assessment variances by different methods.

ELIGIBILITY:
Inclusion Criteria:

* According with ICD-10 criteria of depression;
* Age 16-70;
* Antidepressant and other Psychiatric drugs have not been had two weeks before the trial, or the drugs above had been used but have cleaning period of two weeks;
* Level of education is higher than junior middle school;
* Course of disease is more than two weeks;
* Volunteer to join and Signed the informed consent

Exclusion Criteria:

* Pregnancy or lactation;
* Severe depression or have serious suicidal tendencies
* long distance or other causes who can not adherence to treatment

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
psychological questionnaires | 12 weeks post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Wang, master, Study Chair — Guang'anmen Hospital
Locations (1):
- Guang'anmen Hospital, Beijing, Beijing Municipality, China